CLINICAL TRIAL: NCT04729101
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Vonoprazan (20 mg) and Lansoprazole (30 mg) in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Vonoprazan and Lansoprazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VONO-103
Record Dates: First submitted 2021-01-19; First posted 2021-01-28 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-06

CONDITIONS: Healthy Participants
Keywords: Vonoprazan; Lansoprazole
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (vonoprazan) (Experimental): Participants will be randomized to receive vonoprazan (treatment A) and lansoprazole (treatment B) in a two period sequence, following either treatment sequence AB or BA. There will be a washout period of at least 7 days between Period 1 and Period 2.
  Vonoprazan will be administered via 20 mg oral tablet once daily on Day 1 through to Day 7 in a period, where each period is up to 8 days.
  Interventions: Drug: Vonoprazan
- Treatment B (lansoprazole) (Active Comparator): Participants will be randomized to receive vonoprazan (treatment A) and lansoprazole (treatment B) in a two period sequence, following either treatment sequence AB or BA. There will be a washout period of at least 7 days between Period 1 and Period 2.
  Lansoprazole will be administered via 30 mg oral capsule once daily on Day 1 through to Day 7 in a period, where each period is up to 8 days.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Vonoprazan — Oral tablet
  Arms: Treatment A (vonoprazan)
Drug: Lansoprazole — Oral capsule
  Arms: Treatment B (lansoprazole)

SUMMARY:
To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of vonoprazan (20 mg) and lansoprazole (30 mg) following single (Day 1) and multiple doses (Day 7).

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* Participants must fulfill all the following inclusion criteria to be eligible for participation in the study:

  1. Healthy, adult, male or female 18 - 55 years of age, inclusive, at screening.
  2. Continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on participant self-reporting.
  3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2 at screening.
  4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the principal investigator (PI) or designee.
  5. Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and gamma-glutamyl transferase (GGT) < upper limits of the clinical laboratory reference range (one recheck is permissible).
  6. A female of childbearing potential is either sexually inactive (abstinent as a life style) for 28 days prior to the first dosing and throughout the study or is using one of the following acceptable birth control methods:

     * hormonal oral contraceptives, vaginal ring, transdermal patch, or hormone releasing intrauterine device for at least 3 months prior to the first dosing and with either a physical (e.g., condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study.
     * Depot/implantable hormone (e.g., Depo-Provera®, Implanon®) for at least 3 months prior to the first dosing and throughout the study.

     In addition, female participants of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 28 days after the last dose.
  7. A female of non-childbearing potential has undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

     * hysteroscopic sterilization;
     * bilateral tubal ligation or bilateral salpingectomy;
     * hysterectomy;
     * bilateral oophorectomy;

     or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status.
  8. A non-vasectomized, male participant must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non-vasectomized male).
  9. If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
  10. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

* Participants must not be enrolled in the study if they meet any of the following criteria:

  1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
  2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the principal investigator (PI) or designee.
  3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
  4. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
  5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s), its excipients, related compounds, or lidocaine.
  6. Clinically significant gastrointestinal (GI) disorder (e.g., gastric ulcer (GU), Gastroesophageal reflux disease (GERD), impaction, chronic constipation, inflammatory bowel disease, ischemic colitis, vascular intestinal atherosclerosis, previous bowel resection, bowel obstruction, bariatric surgery, cholecystitis [including history of cholecystectomy], and/or appendectomy).
  7. Positive result for H. pylori breath test at screening.
  8. Had diarrhea or vomiting within 48 hours prior to check-in.
  9. Has nasal abnormalities that could affect pH probe insertion.
  10. Cannot tolerate placement of the pH probe.
  11. Female participants with a positive pregnancy test at screening or check-in or who are lactating.
  12. Positive urine drug or alcohol results at screening or check-in.
  13. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
  14. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
  15. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
  16. Fridericia's correction to the QT interval (QTcF) interval is >460 msec (males) or >470 msec (females) or has electrocardiogram (ECG) findings deemed abnormal with clinical significance by the PI or designee at screening.
  17. Estimated creatinine clearance <80 mL/min at screening.
  18. The participant has serum creatinine >1.22 mg/dL at screening or check-in.
  19. Unable to refrain from or anticipates the use of:

      * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed. After randomization, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee. Topical lidocaine may be administered for pH probe insertion. Hormone replacement therapy will also be allowed.
      * Any drugs known to be significant inducers of CYP3A4/5, CYP1A2, and/or CYP2C19 for 28 days prior to the first dosing and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK / PD interaction with study drug.
  20. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing and throughout the study.
  21. Donation of blood or significant blood loss within 56 days prior to the first dosing.
  22. Plasma donation within 7 days prior to the first dosing.
  23. Participation in another clinical study within 30 days prior to the first dosing. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals, Inc.
Locations (1):
- Celerion, 2420 W Baseline Rd,, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laine L, Sharma P, Mulford DJ, Hunt B, Leifke E, Smith N, Howden CW. Pharmacodynamics and Pharmacokinetics of the Potassium-Competitive Acid Blocker Vonoprazan and the Proton Pump Inhibitor Lansoprazole in US Subjects. Am J Gastroenterol. 2022 Jul 1;117(7):1158-1161. doi: 10.14309/ajg.0000000000001735. Epub 2022 Mar 16. PMID 35294415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 participants were enrolled between January 2021 and June 2021 at a single site in the United States.
Pre-assignment Details: Overall, 164 participants were screened of which 120 were considered screen failures. Eligible participants were randomized to 1 of the 2 treatment sequences in a 1:1 ratio.
Groups:
- First Vonoprazan, Then Lansoprazole (Treatment Sequence AB): Participants received 20 mg vonoprazan (treatment A) as oral tablets once daily (QD) for up to 7 days in Treatment Period 1. Following a 7 day washout period, participants received 30 mg lansoprazole (treatment B) as oral capsules QD for up to 7 days in Treatment Period 2.
- First Lansoprazole, Then Vonoprazan (Treatment Sequence BA): Participants received 30 mg lansoprazole (treatment B) as oral capsules QD for up to 7 days in Treatment Period 1. Following a 7 day washout period, participants received 20 mg vonoprazan (treatment A) as oral tablets QD for up to 7 days in Treatment Period 2.
Period: Overall Study
Arm/Group | First Vonoprazan, Then Lansoprazole (Treatment Sequence AB) | First Lansoprazole, Then Vonoprazan (Treatment Sequence BA)
Started | 23 | 21
Received Treatment | 23 | 21
Completed | 20 | 21
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population - all participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Vonoprazan, Then Lansoprazole (Treatment Sequence AB) | First Lansoprazole, Then Vonoprazan (Treatment Sequence BA) | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.30) | 37.1 (9.99) | 36.1 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 15 | 17 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Black or African American | 3 | 2 | 5
  Native Hawaiian/Pacific Islander | 0 | 1 | 1
  White | 17 | 15 | 32
  White, Asian | 1 | 0 | 1
  White, Black or African American | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Gastric pH >4 Holding Time Ratio (HTR): Percentage of Time Gastric pH Was Above 4 Over a 24-hour Monitoring Period Following Study Drug Administration
Description: Calculated as: Time pH >4*100/total actual monitoring period time. Gastric pH was measured continuously over a 24-hour period on Days 1 and 7 of Periods 1 and 2, using a pH and pressure sensitive probe and ambulatory pH recording system. A pH recording was taken every second.
Time Frame: Day 1 and Day 7 of each treatment period
Population: Pharmacodynamic (PD) Population - all participants who received at least one dose of the study drug and had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Vonoprazan: Participants received 20 mg vonoprazan (treatment A) as oral tablets QD for up to 7 days in Treatment Period 1 or Treatment Period 2.
- Lansoprazole: Participants received 30 mg lansoprazole (treatment B) as oral capsules QD for up to 7 days in Treatment Period 1 or Treatment Period 2.
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 41
percentage of time
  Day 1 | 62.40 (23.351) | 22.61 (17.309)
  Day 7: number analyzed (Participants) | 40 | 38
  Day 7 | 87.81 (15.708) | 42.32 (25.597)
Statistical Analysis 1: Comparison: Vonoprazan vs Lansoprazole; Vonoprazan versus lansoprazole on Day 1 of each treatment period; Test type: Other — Additional statistics were descriptive in nature; Least-squares mean difference = 38.98, 95% CI 2-sided [31.94 to 46.02]
Statistical Analysis 2: Comparison: Vonoprazan vs Lansoprazole; Vonoprazan versus lansoprazole on Day 7 of each treatment period; Test type: Other — Additional statistics were descriptive in nature; Least-squares mean difference = 44.62, 95% CI 2-sided [37.55 to 51.69]

2. Primary Outcome: Mean Gastric pH Over a 24-hour Monitoring Period Following Study Drug Administration (pH0-24)
Description: The average gastric pH was a measure of the immediate effect on gastric pH and the duration of effect on gastric pH. Gastric pH was measured continuously over a 24-hour period on Days 1 and 7 of Periods 1 and 2, using a pH and pressure sensitive probe and ambulatory pH recording system. A pH recording was taken every second. The pH scale ranges from 0 to 14 with values below 7 being more acidic and values above 7 being more basic. Normal gastric pH is between 1.5 and 3.5.
Time Frame: Day 1 and Day 7 of each treatment period
Population: PD Population - all participants who received at least one dose of the study drug and had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 41
pH
  Day 1 | 4.606 (1.0852) | 2.848 (0.79923)
  Day 7: number analyzed (Participants) | 40 | 38
  Day 7 | 5.903 (0.84900) | 3.783 (1.2000)
Statistical Analysis 1: Comparison: Vonoprazan vs Lansoprazole; Vonoprazan versus lansoprazole on Day 1 of each treatment period; Test type: Other — Additional statistics were descriptive in nature; Least-squares mean difference = 1.72, 95% CI 2-sided [1.40 to 2.04]
Statistical Analysis 2: Comparison: Vonoprazan vs Lansoprazole; Vonoprazan versus lansoprazole on Day 7 of each treatment period; Test type: Other — Additional statistics were descriptive in nature; Least-squares mean difference = 2.09, 95% CI 2-sided [1.74 to 2.44]

3. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to the 24-Hour Time Point (AUC0-24)
Description: Calculated using the Linear Trapezoidal with Linear Interpolation Method. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 1: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (Pharmacokinetics [PK]) - all participants with an evaluable AUC0-24 profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 41
ng*hr/mL | 200.6 (80.954) | 2677 (1357.1)

4. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf)
Description: Calculated as the area under the concentration-time curve, from time 0 to the last observed non-zero concentration (AUC0-t) + (Clast/Kel) where Clast is the last observed/measured concentration and Kel is the apparent first-order terminal elimination rate constant. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 1: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable AUC0-inf profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 39 | 41
ng*hr/mL | 229.5 (98.841) | 2679 (1361.0)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was taken directly from bioanalytical data. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 1: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable Cmax profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 41
ng/mL | 21.79 (8.3296) | 1110 (411.88)

6. Primary Outcome: Time to Reach Cmax (Tmax)
Description: Taken from the clinical database as the difference in the time of administration and the time of the blood draw which was associated with the Cmax. If the maximum value occurred at more than one time point, Tmax was defined as the first time point with this value. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 1: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable Tmax profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Median (Full Range); unit: hr
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 41
hr | 2.005 [1.00 to 5.01] | 1.499 [0.79 to 4.00]

7. Primary Outcome: Area Under the Concentration-Time Curve During a Dosing Interval (AUCtau) at Steady State (ss)
Description: as for outcome 3
Time Frame: Day 7: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable AUCtau profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 38
ng*hr/mL | 261.4 (104.18) | 3246 (2396.4)

8. Primary Outcome: Cmax at Steady State (Cmax,ss)
Description: Cmax,ss was taken directly from bioanalytical data. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 7: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable Cmax,ss profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 38
ng/mL | 27.39 (9.9928) | 1164 (506.53)

9. Primary Outcome: Tmax at Steady State (Tmax,ss)
Description: Taken from the clinical database as the difference in the time of administration and the time of the blood draw which was associated with the Cmax,ss. The analyses of vonoprazan and lansoprazole in plasma samples was performed using validated liquid chromatography-mass spectrometry/mass spectrometry methods.
Time Frame: Day 7: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 9, 10, 12, 13, 16, and 24 hours postdose
Population: PD Population (PK) - all participants with an evaluable PK profile who received at least one dose of the study drug had sufficient predose and postdose pH measurements and absence of major protocol violations.
Measure: Median (Full Range); unit: hr
Arm/Group | Vonoprazan | Lansoprazole
Number analyzed (Participants) | 40 | 38
hr | 2.005 [1.53 to 5.00] | 1.510 [0.75 to 4.02]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 35
Description: The adverse events reported are treatment-emergent adverse events which were defined as any event that occurred after the first dose of study drug or any event at baseline that worsened in either intensity or frequency after the first dose of study drug. The analysis population was the safety population which included all participants who received at least one dose of the study drug.
Arm/Group | Vonoprazan | Lansoprazole
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 9/44 | 17/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan (N=44) | Lansoprazole (N=43)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Nodule (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Vaginitis gardnerella (Infections and infestations) | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04729101/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04729101/SAP_001.pdf